CLINICAL TRIAL: NCT06414707
Title: Efficacy of Vonoprazan Versus Proton Pump Inhibitors in Combination With Antibiotics as a Triple Therapy for Eradication of Clarithromycin Resistant Strain of Helicobacter Pylori
Brief Title: Efficacy of Vonoprazan in Eradication of Resistant Strain of Helicobacter Pylori
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R288/2023
Record Dates: First submitted 2024-04-06; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Levofloxacin; Ofloxacin; Pantoprazole

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial included two groups of Egyptian patients diagnosed with dyspepsia related to Clarithromycin-resistant strains of H.pylori.
  * Group (1) ( Vonoprazan Group) included 160 patients received Vonoprazan 20 mg oral once daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for two weeks.
  * Group (2)(Pantoprazole Group) included 160 patients received Pantoprazole 40 mg oral twice daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for 14 days.
  All cases were diagnosed with H. Pylori resistant infection after clarithromycin based treatment regimen for H. pylori confirmed with persistent positive test of fecal H. pylori Ag before the starting of the study.
  All patients of the two groups were followed up for persistence of infection 8-weeks following the end of therapy by testing fecal H. pylori Ag.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vonoprazan Group (Active Comparator): included 160 patients received Vonoprazan 20 mg oral once daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for two weeks.
  Interventions: Drug: Vonoprazan, Amoxicillin and Levofloxacin
- Pantoprazole Group (Active Comparator): included 160 patients received Pantoprazole 40 mg oral twice daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for 14 days
  Interventions: Drug: Pantoprazole 40mg, Amoxicillin and Levofloxacin

INTERVENTIONS:
Drug: Vonoprazan, Amoxicillin and Levofloxacin — Group (1) included 160 patients received Vonoprazan 20 mg oral once daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for 14 days.
  Other Names: Vonaspire 20 mg; Amoxil 1 gm; Tavanic 500 mg
  Arms: Vonoprazan Group
Drug: Pantoprazole 40mg, Amoxicillin and Levofloxacin — Group (2) included 160 patients received Pantoprazole 40 mg oral twice daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for 14 days.
  Other Names: controloc 40 mg; Amoxil 1 gm; Tavanic 500 mg
  Arms: Pantoprazole Group

SUMMARY:
The goal of this Randomized controlled trial is to assessment Efficacy of Vonoprazan versus Proton Pump Inhibitors in Combination with Antibiotics as a triple Therapy for Eradication of Clarithromycin Resistant Strain of Helicobacter Pylori (H. pylori).

This randomized controlled study was performed on 2 groups of Egyptian patients diagnosed with dyspepsia; group (1) included 160 patients received Vonoprazan 20 mg oral once daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for 14 days and group (2) included 160 patients received Pantoprazole 40 mg oral twice daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for 14 days. All patients of the two groups were followed up for persistence of infection 8 weeks after the end of treatment by testing fecal H. pylori antigen (Ag).

DETAILED DESCRIPTION:
This randomized controlled trial included two groups of Egyptian patients diagnosed with dyspepsia related to Clarithromycin-resistant strains of H.pylori.

* Group (1) included 160 patients received Vonoprazan 20 mg oral once daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for two weeks.
* Group (2) included 160 patients received Pantoprazole 40 mg oral twice daily + Levofloxacin 500 mg oral once daily + Amoxicillin 1 gm oral twice daily for 14 days.

The included cases were collected from gastroenterology outpatient clinic and inpatient department at Ain shams University hospital between October 2023 and April 2024.

The work had been conducted after the scientific ethics committee approval and after obtaining an informed consent from all the included cases.

All cases were diagnosed with H. Pylori resistant infection after clarithromycin based treatment regimen for H. pylori confirmed with persistent positive test of fecal H. pylori Ag before the starting of the study.

All patients of the two groups were followed up for persistence of infection 8-weeks following the end of therapy by testing fecal H. pylori Ag. And the study end-points were compliance failure or gastrointestinal bleeding.

Each participant had been exposed to comprehensive taking of history, full physical assessment, full laboratory examination including (CBC, liver profile (ALT, AST), kidney functions test (S. creat), fecal H. pylori Ag testing before the starting of the trial and another stool sample were taken after termination of treatment by 8 weeks for evaluating of the eradication of H. pylori infection and pelvi-abdominal U/S was done for all patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with dyspepsia related to Clarithromycin-resistant strains of H.pylori. All cases were diagnosed with H. Pylori resistant infection after clarithromycin based treatment regimen for H. pylori confirmed with persistent positive test of fecal H. pylori Ag before the starting of the study.
* Must be able to swallow tablets.

Exclusion Criteria:

* Cases with drug allergy from drugs included in the study.
* those having inflammatory-bowel diseases.
* those with malabsorption syndrome.
* those having gastroenterology malignancy.
* patients on immunotherapy.
* HIV patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Assessment the fecal H.Pylori Ag after receiving Vonoprazan in combination with antibiotics as a triple therapy in patients with Clarithromycin-resistant strain of H.Pylori infection. | All patients of the two groups were followed up for 2 months.
  comparison between the efficiency of Vonoprazan and Pantoprazole in eradication of Clarithromycin-resistant strain of H.Pylori.

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Elfors, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No